CLINICAL TRIAL: NCT01669174
Title: A Randomized, Double Blind, Placebo Controlled, Multi-centre Study to Asses the Pharmacodynamics, Pharmacokinetics, Safety and Tolerability of BYM338 in Chronic Obstructive Pulmonary Disease Patients With Cachexia
Brief Title: BYM338 in Chronic Obstructive Pulmonary Disease (COPD) Patients With Cachexia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: CBYM338X2204; 2011-000461-12
Record Dates: First submitted 2012-03-01; First posted 2012-08-20 (Estimated); Results first posted 2016-05-03 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-04

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD) With Cachexia
Keywords: Chronic Obstructive Pulmonary Disease; COPD; cachexia; muscle wasting
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Cachexia; Muscular Atrophy | interventions — bimagrumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BYM338 (Experimental)
  Interventions: Drug: BYM338
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo
  Arms: Placebo
Drug: BYM338 — BYM338
  Arms: BYM338

SUMMARY:
This study will assess the pharmacodynamics, pharmacokinetics, safety and tolerability of BYM338 in patients with COPD and cachexia. The primary outcome will be a change in thigh muscle volume compared to placebo. The study will last for approximately 24 weeks.

ELIGIBILITY:
Inclusion criteria:

* Written informed consent must be obtained before any assessment is performed.
* Males and females ages 40 to 80 years
* Smoking history of at least 10 pack-years
* Diagnosis of COPD according to GOLD guidelines (GOLD, 2010), with a post-bronchodilator FEV¬1 < 80% predicted and FEV1/FVC ratio < 0.70
* BMI <20 kg/m2 or skeletal muscle mass index by DXA < 7.25 kg/m2 for men or <5.45 kg/m2 for women.
* In general stable health, including managed COPD, by past medical history, physical examination, vital signs at baseline as determined by the investigator.

Exclusion criteria:

* Patients with MRC dyspnoea grade 5 (i.e. patients too breathless to leave the house or breathless when dressing)
* Plans for lung transplantation or lung reduction surgery within four months of enrollment
* Patients participating in a formal pulmonary rehabilitation program within 3 months of dosing
* History of malignancy of any organ system (other than excised non-melanomatous carcinoma of the skin), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
* Diseases other than cancer known to cause cachexia or muscle atrophy, including but not limited to congestive heart failure of any stage, chronic kidney disease (estimated GFR < 30 mL/min using the MDRD equation), rheumatoid arthritis, primary myopathy, stroke, HIV infection, tuberculosis or other chronic infection, uncontrolled diabetes mellitus, etc.
* Inflammatory bowel disease, celiac disease, short bowel syndrome, pancreatic insufficiency
* Use of any prescription drugs known to affect muscle mass, including androgen supplements, anti-androgens (such as LHRH agonists), anti-estrogens (tamoxifen, etc.) recombinant human growth hormone (rhGH), insulin, oral beta agonists, megestrol acetate, dronabinol, metformin, etc.
* Hemoglobin concentration below 11.0 g/dL at screening.
* Liver disease or liver injury.
* Use of other investigational drugs at the time of enrollment, or within 30 days and for any other limitation of participation in an investigational trial based on local regulations.
* Women of child-bearing potential.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2012-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (9):
- United States (5):
  - Novartis Investigative Site, Torrance, California
  - Novartis Investigative Site, Savannah, Georgia
  - Novartis Investigative Site, Normal, Illinois
  - Novartis Investigative Site, Missoula, Montana
  - Novartis Investigative Site, Spartanburg, South Carolina
- Novartis Investigative Site, Maastricht, Netherlands
- United Kingdom (3):
  - Novartis Investigative Site, Leicester
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Machester

REFERENCES:
- [Derived] Polkey MI, Praestgaard J, Berwick A, Franssen FME, Singh D, Steiner MC, Casaburi R, Tillmann HC, Lach-Trifilieff E, Roubenoff R, Rooks DS. Activin Type II Receptor Blockade for Treatment of Muscle Depletion in Chronic Obstructive Pulmonary Disease. A Randomized Trial. Am J Respir Crit Care Med. 2019 Feb 1;199(3):313-320. doi: 10.1164/rccm.201802-0286OC. PMID 30095981

RESULTS

PARTICIPANT FLOW:
Groups:
- BYM338: 30 mg/kg
- Placebo: Placebo to BYM338 30mg/kg
Period: Overall Study
Arm/Group | BYM338 | Placebo
Started | 33 | 34
Completed | 27 | 28
Not Completed | 6 | 6
Not completed — Subject withdrew consent | 2 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Adverse Event | 2 | 2
Not completed — Administrative problems | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BYM338 | Placebo | Total
Number analyzed (Participants) | 33 | 34 | 67
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.5 (5.93) | 63.1 (7.51) | 63.7 (6.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 18 | 34
  Male | 17 | 16 | 33

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline of Thigh Muscle Volume (TMV) by MRI Scan at Week 4, 8, 16, and 24
Description: Thigh Muscle Volume (TMV) change was evaluated by a responder analysis. Patients whose loss of muscle TMV by MRI was no more than or equal to 2% at Week 4,8,16 and 24 was considered responders.
Time Frame: Baseline, Weeks 4, 8, 16, 24
Population: Pharmacodynamics (PD) analysis set: Patients with evaluable PD parameter data. However, for a given time frame, analyzed participants had values at both baseline and the corresponding time frame.
Measure: Mean (Standard Deviation); unit: Percentage Change of TMV
Arm/Group | BYM338 | Placebo
Number analyzed (Participants) | 33 | 34
Percentage Change of TMV
  Week 4 Day 29 (n=30,31) | 5.87 (3.413) | 0.02 (3.261)
  Week 8 Day 57 (n=27,27) | 7.01 (3.707) | -0.65 (2.752)
  Week 16 Day 113 (27,28) | 7.84 (5.052) | -0.88 (4.471)
  End of Study, week 24 (n=27,28) | 5.04 (4.872) | -1.31 (4.282)
Statistical Analysis 1: Comparison: BYM338 vs Placebo; Week 4; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Net) = 106.10, 90% CI 2-sided [104.64 to 107.58]
Statistical Analysis 2: Comparison: BYM338 vs Placebo; Week 8; Test type: Superiority or Other; p < 0.001, ANCOVA; Median Difference (Net) = 107.75, 90% CI 2-sided [106.18 to 109.35]
Statistical Analysis 3: Comparison: BYM338 vs Placebo; Week 16; Test type: Superiority or Other; p < 0.001, ANCOVA; Median Difference (Net) = 108.63, 90% CI 2-sided [106.31 to 111.00]
Statistical Analysis 4: Comparison: BYM338 vs Placebo; Week 24; Test type: Superiority or Other; p < 0.001, ANCOVA; Median Difference (Net) = 106.63, 90% CI 2-sided [104.39 to 108.93]

2. Secondary Outcome: Change in 6 Minute Walk Distance Compared to Placebo
Description: Practical simple test that requires a 100-ft hallway but no exercise quipment or advanced training for technicians. Walking is an activity performed daily by all but the most severely impaired patients. This test measures the distance that a patient can quickly walk on a flat, hard surface in a period of 6 minutes (the 6MWD)
Time Frame: Baseline, Weeks 4, 8, 16, 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: meter
Arm/Group | BYM338 | Placebo
Number analyzed (Participants) | 33 | 34
meter
  Week 4 Day 29 (n=30,32) | 364.6 (85.45) | 388.5 (100.22)
  Week 8 Day 57 (n=27,29) | 373.9 (101.42) | 387.4 (99.73)
  Week 12 Day 85 (n=27,28) | 383.0 (84.63) | 385.6 (107.62)
  Week 16 Day 113 (n=25,28) | 379.7 (83.78) | 352.9 (104.01)
  End of Study week 24 (n=27, 28) | 374.9 (98.29) | 378.8 (81.50)

3. Secondary Outcome: Maximum Observed Serum Concentration (Cmax)
Description: The observed maximum plasma concentration following drug administration
Time Frame: 0 hour, 2 hour, Day 8, 15, 29, 57, 71, 85, 99, 113, 127, 168 post dose
Population: Pharmacokinetics (PK) analysis set: Patients with evaluable PK data.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | BYM338
Number analyzed (Participants) | 33
ug/mL
  Cmax dose 1 (n=31) | 614 (143)
  Cmax dose 2 (n=26) | 580 (121)

4. Secondary Outcome: Time to Reach the Maximum Concentration After Drug Administration (Tmax)
Description: The time to reach the maximum concentration after drug administration
Time Frame: 24 weeks
Population: Pharmacokinetics (PK) analysis set: Patients with evaluable PK data.
Measure: Median (Full Range); unit: hr
Arm/Group | BYM338
Number analyzed (Participants) | 33
hr
  Tmax dose 1 (n=31) | 2.22 (NA) [2.02 to 3.17]
  Tmax dose 2 (n=26) | 2.23 (NA) [1.97 to 3.20]

5. Secondary Outcome: AUC0-56 and AUClast
Description: AUC0-56, the area under the serum concentration-time curve from the time zero to the end of the dosing interval, day 56. AUC0-56 was analyzed for dose 1 and 2. AUClast is from time zero to the last quantifiable concentration. AUClast was analyzed for dose 2 only.
Time Frame: 0 hour, 2 hour, Day 8, 15, 29, 57, 71, 85, 99, 113, 127, 168 post dose
Population: Pharmacokinetics (PK) analysis set: Patients with evaluable PK data.
Measure: Mean (Standard Deviation); unit: day*ug/mL
Arm/Group | BYM338
Number analyzed (Participants) | 33
day*ug/mL
  AUC0-56 dose 1 (n=26) | 4540 (897)
  AUC0-56 dose 2 (n=25) | 5790 (1300)
  AUClast dose 2 (n=25) | 7480 (2080)

ADVERSE EVENTS:
Groups:
- BYM338 30mg/kg: BYM338 30mg/kg
Arm/Group | BYM338 30mg/kg | Placebo
Serious Adverse Events (participants affected / at risk) | 4/33 | 3/34
Other Adverse Events (participants affected / at risk) | 31/33 | 30/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BYM338 30mg/kg (N=33) | Placebo (N=34)
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 1
Postoperative wound infection (Infections and infestations) | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BYM338 30mg/kg (N=33) | Placebo (N=34)
Atrial fibrillation (Cardiac disorders) | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 7 | 3
Dyspepsia (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 1
Fatigue (General disorders) | 2 | 3
Feeling abnormal (General disorders) | 4 | 3
Feeling cold (General disorders) | 2 | 0
Influenza like illness (General disorders) | 2 | 0
Oedema peripheral (General disorders) | 0 | 2
Pain (General disorders) | 0 | 2
Gastroenteritis (Infections and infestations) | 2 | 1
Nasopharyngitis (Infections and infestations) | 4 | 0
Pneumonia (Infections and infestations) | 1 | 2
Rash pustular (Infections and infestations) | 3 | 2
Sinusitis (Infections and infestations) | 3 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 4
Contusion (Injury, poisoning and procedural complications) | 2 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 2
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 2
Alanine aminotransferase increased (Investigations) | 3 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 0
Blood alkaline phosphatase increased (Investigations) | 2 | 0
Blood creatine phosphokinase increased (Investigations) | 2 | 2
Blood glucose increased (Investigations) | 2 | 1
Gamma-glutamyltransferase increased (Investigations) | 3 | 0
Haemoglobin urine present (Investigations) | 2 | 2
Urine leukocyte esterase positive (Investigations) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 4
Joint lock (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 26 | 16
Muscle tightness (Musculoskeletal and connective tissue disorders) | 18 | 5
Muscle twitching (Musculoskeletal and connective tissue disorders) | 15 | 9
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 3 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 6
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 7
Dizziness (Nervous system disorders) | 3 | 3
Headache (Nervous system disorders) | 3 | 8
Paraesthesia (Nervous system disorders) | 3 | 1
Anxiety (Psychiatric disorders) | 0 | 2
Depression (Psychiatric disorders) | 1 | 3
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 16 | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acne (Skin and subcutaneous tissue disorders) | 3 | 1
Blister (Skin and subcutaneous tissue disorders) | 2 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 2
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 | 2
Erythema (Skin and subcutaneous tissue disorders) | 4 | 4
Papule (Skin and subcutaneous tissue disorders) | 2 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 7
Rash (Skin and subcutaneous tissue disorders) | 0 | 2
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 3
Haematoma (Vascular disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety